CLINICAL TRIAL: NCT00433602
Title: TEACH Survey (Thrombo-Embolism And Chemotherapy) A Prospective Survey on the Incidence of Venous Thromboembolic Events During Chemotherapy for Solid Tumors
Brief Title: Incidence of Blood Clots in Patients Undergoing Chemotherapy for Solid Tumors
Status: Completed | Type: Observational
Sponsor: European Organisation for Research and Treatment of Cancer - EORTC (Network)
Responsible Party: Sponsor
Other Study IDs: EORTC-90051; EORTC-90051; SANOFI-AVENTIS-EORTC-90051
Record Dates: First submitted 2007-02-08; First posted 2007-02-12 (Estimated); Last update posted 2013-06-12 (Estimated); Status verified 2013-06

CONDITIONS: Breast Cancer; Colorectal Cancer; Gastric Cancer; Lung Cancer; Ovarian Cancer; Pancreatic Cancer; Prostate Cancer; Thromboembolism
Keywords: thromboembolism; recurrent breast cancer; stage IV breast cancer; recurrent colon cancer; stage I colon cancer; stage II colon cancer; stage III colon cancer; stage IV colon cancer; recurrent rectal cancer; stage I rectal cancer; stage II rectal cancer; stage III rectal cancer; stage IV rectal cancer; recurrent gastric cancer; stage I gastric cancer; stage II gastric cancer; stage III gastric cancer; stage IV gastric cancer; recurrent non-small cell lung cancer; stage I non-small cell lung cancer; stage II non-small cell lung cancer; stage IIIA non-small cell lung cancer; stage IIIB non-small cell lung cancer; stage IV non-small cell lung cancer; recurrent small cell lung cancer; recurrent ovarian epithelial cancer; stage I ovarian epithelial cancer; stage II ovarian epithelial cancer; stage III ovarian epithelial cancer; stage IV ovarian epithelial cancer; recurrent ovarian germ cell tumor; stage I ovarian germ cell tumor; stage II ovarian germ cell tumor; stage III ovarian germ cell tumor; stage IV ovarian germ cell tumor; ovarian sarcoma; ovarian stromal cancer; recurrent pancreatic cancer; stage I pancreatic cancer; stage II pancreatic cancer; stage III pancreatic cancer; stage IV pancreatic cancer; recurrent prostate cancer; stage III prostate cancer; stage IV prostate cancer; extensive stage small cell lung cancer; limited stage small cell lung cancer; stage IIB prostate cancer; stage IIA prostate cancer; male breast cancer
MeSH Terms: conditions — Breast Neoplasms; Colorectal Neoplasms; Stomach Neoplasms; Lung Neoplasms; Ovarian Neoplasms; Pancreatic Neoplasms; Prostatic Neoplasms; Thromboembolism; Colonic Neoplasms; Rectal Neoplasms; Carcinoma, Non-Small-Cell Lung; Small Cell Lung Carcinoma; Carcinoma, Ovarian Epithelial; Breast Neoplasms, Male | interventions — Watchful Waiting; High-Energy Shock Waves

INTERVENTIONS:
Other: clinical observation
Procedure: management of therapy complications
Procedure: ultrasound imaging

SUMMARY:
RATIONALE: Chemotherapy may cause blood clots to form in the thigh, leg, and lung. This study may help doctors understand how often blood clots occur in patients undergoing chemotherapy.

PURPOSE: This clinical trial is studying how often blood clots occur in patients undergoing chemotherapy for solid tumors, including colorectal cancer, stomach cancer, lung cancer, ovarian cancer, pancreatic cancer, prostate cancer, or metastatic breast cancer

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the incidence of venous thromboembolic events (i.e., deep vein thrombosis and/or pulmonary embolism) in patients undergoing chemotherapy for solid tumors.

OUTLINE: This is a prospective, multicenter survey.

Patients undergo observation beginning on day 1 of chemotherapy and continuing for up to 3 months in the absence of symptomatic, confirmed deep vein thrombosis or pulmonary embolism; use of anticoagulant therapy for more than 5 days as curative treatment; or initiation of thromboprophylaxis for any reason. Patients undergo bilateral compression ultrasound of the lower limbs at baseline and at 3 months (or at an earlier timepoint, if indicated).

PROJECTED ACCRUAL: A total of 2,000 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Cytologically or histologically confirmed diagnosis of 1 of the following:

  * Metastatic breast cancer
  * Colorectal cancer
  * Gastric cancer
  * Lung cancer
  * Ovarian cancer
  * Pancreatic cancer
  * Hormone-refractory prostate cancer
* Scheduled to undergo chemotherapy for ≥ 3 months

  * Chemotherapy for colorectal, gastric, lung, ovarian, or pancreatic cancer may be administered in the neoadjuvant, adjuvant, or palliative setting
* History of deep vein thrombosis or pulmonary embolism allowed if treatment and secondary prevention of the last episode was completed prior to study entry

  * Negative baseline bilateral compression ultrasonography

PATIENT CHARACTERISTICS:

* Life expectancy > 3 months

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* More than 6 weeks since prior chemotherapy*

  * Hormonal therapy alone is not considered chemotherapy
* More than 4 weeks since prior major surgery, including surgery for cancer

  * Minor surgery (e.g., implant of a port-a-cath) within the past 4 weeks allowed
* No concurrent major surgery, including surgery for cancer, during the observation period
* Radiotherapy before or during the observation period allowed
* Concurrent chemotherapy* in combination with additional hormonal therapy allowed
* Concurrent treatment (with the exception of antithrombotic therapy) in any other clinical trial allowed
* No concurrent or scheduled use of thromboprophylaxis or any anticoagulant therapy, including any of the following:

  * Parenteral anticoagulants (e.g., heparin, low molecular-weight heparin, or other agents, such as fondaparinux or bivalirudin)
  * Oral anticoagulants (e.g., vitamin K antagonists)
  * Thrombolytic agents

    * Chronic treatment with antiplatelet agents, such as low-dose aspirin (≤ 300 mg/day) or clopidogrel allowed NOTE: *Chemotherapy is defined as treatment with any antineoplastic agent, including biologicals

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2006-11; Primary Completion 2007-03 (Actual)

PRIMARY OUTCOMES:
Incidence of asymptomatic proximal deep vein thrombosis (DVT) of the lower limbs as assessed by bilateral compression ultrasound at baseline and at 3 months
Incidence of symptomatic, proximal and/or distal DVT of the lower limbs as assessed by clinical diagnosis and compression ultrasound within 72 hours of detection of symptoms (during the 3-month observation period)
Incidence of symptomatic pulmonary embolism as assessed by ventilation/perfusion lung scan, pulmonary angiogram, or CT lung scan within 72 hours of detection of symptoms or during autopsy (during the 3-month observation period)

CONTACTS AND LOCATIONS:
Overall Officials: Hans-Martin Otten, MD, Study Chair — Slotervaart Ziekenhuis; Ullrich Bethe, MD, Study Chair — European Organisation for Research and Treatment of Cancer - EORTC
Locations (1):
- Slotervaart Ziekenhuis, Amsterdam, Netherlands